CLINICAL TRIAL: NCT01685047
Title: A Clinical Evaluation of ST Changes in a Group of Patients Having Ventricular Arrhythmias
Acronym: inSighT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-12-014-ID-HV
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Ventricular Arrhythmias; ST Segment Changes
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this investigation is to determine the prevalence of device-recorded ST segment changes occurring before appropriate Implantable Cardiac Defibrillator (ICD) therapies (ATP or Shock) and to define their temporal relationship to ventricular arrhythmias.

DETAILED DESCRIPTION:
Sudden cardiac death due to cardiac arrhythmia is a devastating and unpredictable complication of coronary artery disease.

Implantation of automatic implantable cardioverter defibrillators (ICD) is a well established therapy for the treatment and prevention of sudden cardiac death. Evidence for the use of these devices has been provided by a number of landmark clinical trials over the last 16 years.

Reduction in ischemia can be achieved by coronary artery revascularization but in many patients may occur a gradual progression to recurrence of ischemia resulting in further life threatening arrhythmias. It is reasonable to assume that unchecked progression of ischemic heart disease may result in increased mortality in ICD patients. It has been shown that the long term mortality risk for ICD patients can be linked to the time since the last coronary revascularization procedure. Both MADIT-II and Sudden Cardiac Death in Heart Failure trial (SCD-HeFT) showed that patients receiving inappropriate ICD therapy have an increased risk of death. It has been speculated that this may be due to progression of the disease and recurrent ischemia.

A feature available in some ICDs manufactured by St Jude medical enables the constant beat to beat monitoring of the intra-cardiac ST segment using the implanted ICD leads. Similar systems have demonstrated this approach to be a reliable method of identifying ischemic events. However, the predictive value of the ST monitoring feature in identifying pending arrhythmic events has yet to be established. Prediction of worsening ischemia could play an important part in allowing physicians to identify ICD patients with greater mortality risk and allow them the time to personalize patient therapy in order to reduce that risk.

ELIGIBILITY:
Inclusion Criteria:

* The patient is implanted with an St Jude Medical (SJM) ICD with ST Monitoring and ShockGuard™ features (and remote care feature in case Merlin.net will be used)
* The patient, in the opinion of the investigator, will not require ventricular pacing for more than 20% of the time.
* The patient, in the opinion of the investigator, has or is at high risk of Coronary Artery Disease (CAD).
* The patient is ≥ 18 years of age.
* The patient is able to provide written Informed Consent prior to any investigational related procedure.

Exclusion Criteria:

* The patient has longstanding persistent Atrial Fibrillation (AF) /Atrial Flutter (AFl) or permanent AF/AFl
* The patient has documented complete heart block.
* The patient is known to have uncontrolled ventricular bigeminy or trigeminy (PVCs on regular basis).
* The patient has severe Left Ventricular Hypertrophy resulting in interventricular conduction defect (IVCD).
* The patient has intermittent bundle branch blocks (BBB).
* The patient is unable to comply with the follow up schedule.
* The patient is participating in another investigational device or drug investigation.
* The patient is pregnant or is planning to become pregnant during the duration of the investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient is implanted with SJM ICD and has or is at high risk of CAD
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes SPERZEL, MD, Principal Investigator — Kerckhoff Klinik, Bad Nauheim Germany
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Population: Patients implanted with a St. Jude Medical ICD device with ST monitoring and ShockGuard feature, a right ventricular lead and, when applicable, a right atrial lead, were eligible for this investigation.
Period: Overall Study
Arm/Group | Patient Population
Started | 481 (481 subjects signed the consent. 1 subject was withdrawn prior to the baseline visit.)
Completed | 396
Not Completed | 85
Not completed — Withdrawal by Subject | 20
Not completed — Death | 26
Not completed — Lost to Follow-up | 8
Not completed — Physician Decision | 25
Not completed — Adverse Event | 5
Not completed — patient withdrawn by sponsor | 1

BASELINE CHARACTERISTICS:
Population: A total of 481 subjects were enrolled. However, 1 subject was withdrawn immediately after enrollment because this subject was not implanted with the study required device. Therefore, the total number of baseline participants (480) is discrepant to the number of participants started (481).
Arm/Group | Patient Population
Number analyzed (Participants) | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.95 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 400
Indication for Implant [Number; unit: participants]
  Primary prevention | 296
  Secondary prevention | 184
Medical History [Number; unit: participants]
  Arrhythmogenic RV cardiomyopathy | 3
  Diabetic cardiomyopathy | 3
  Dilated cardiomyopathy | 93
  Hypertrophic cardiomyopathy | 9
  Inschemic cardiomyopathy | 366
  Non Ischemic cardiomyopathy | 12
  Obesity associated cardiomyopathy | 1
  Other | 23
Atrial Arrhythmia history [Number; unit: participants]
  Atrial Fibrillation | 76
  Atrial Flutter | 14
Ventricular Arrhythmia history [Number; unit: participants]
  Premature ventricular contractions | 27
  Monomorphic ventricular tachycardia | 107
  Ventricular fibrillation | 79
  Polymorphic ventricular tachycardia | 10
  Other | 23

OUTCOME MEASURES:

1. Primary Outcome: Among Patients With an Appropriate ICD Therapy (Shock or ATP) for Ventricular Tachycardia or Fibrillation, the Number of Patients Who Have Characterized ST Segment Changes From Baseline Prior to the Therapy Was Calculated.
Time Frame: Until the end of follow up period
Population: The other subjects enrolled in this study had no treated VT/VF events.
Measure: Number; unit: participants
Units Other Than Participants: VT/VF events
Arm/Group | Patient Population
Number analyzed (Participants) | 117
Number analyzed (VT/VF events) | 245
participants | 56
Statistical Analysis 1: Comparison: Patient Population; There were no formal pre-specified statistical hypotheses for the endpoints of the study due to the exploratory nature of this study. Some data was excluded from the primary analysis. All device detections resulting in therapy have been reviewed for appropriateness of the therapy. VT/VF therapy delivered from the device as a result of a non-ventricular arrhythmia or as a result of oversensing by the device has not been included in the primary data analysis; Test type: Other — There were no formal pre-specified statistical hypotheses for the endpoints of the study due to the exploratory nature of this study. Datasets (Device info at Baseline versus 15 minutes prior to the event) were compared using a 2-sided t-test; p < 0.05, t-test, 2 sided — All events with p <0.05 were visually inspected to confirm they were evaluable; additional criteria for exclusion from further analysis included inappropriate therapy, aberrant conduction, and occurrence of VT/VF within 24h prior to the event

ADVERSE EVENTS:
Time Frame: Safety surveillance and reporting started as soon as the subject was enrolled until study conclusion. All patients were followed up until the last patient had performed his/her 12 month follow up visit, therefore, no fixed period is available per patient. The study (and follow up period) ended for all patients 26AUG2016.
Arm/Group | Patient Population
Serious Adverse Events (participants affected / at risk) | 147/481
Other Adverse Events (participants affected / at risk) | 57/481
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Population (N=481)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 29 (37)
Cardiac arrest (Cardiac disorders) | 1 (1)
Component failure (Injury, poisoning and procedural complications) | 4 (4) — Device component failure
Death - Cardiovascular related (Cardiac disorders) | 3 (3)
Death - Non cardiovascular related (General disorders) | 3 (3)
Death - Unknown (General disorders) | 5 (5)
Drug Reaction (Injury, poisoning and procedural complications) | 1 (1)
Exacerbation of Heart failure (Cardiac disorders) | 23 (33)
Gastro-enteritis (Gastrointestinal disorders) | 1 (1)
Inappropriate high voltage therapy (Injury, poisoning and procedural complications) | 7 (7)
Infection related to system and/or procedure (Infections and infestations) | 3 (3)
Ischemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Lead dislodgement or migration (Injury, poisoning and procedural complications) | 5 (5)
Inappropriate device function (Surgical and medical procedures) | 1 (1)
Myocardial infarction (Cardiac disorders) | 6 (7)
Other cardiovascular related event (Vascular disorders) | 30 (35)
Other non cardiovascular (Surgical and medical procedures) | 61 (71)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Thromboemboli (Blood and lymphatic system disorders) | 1 (1)
Transient Ischemic Attack (Blood and lymphatic system disorders) | 1 (1)
Veinthrombosis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Population (N=481)
Arrhythmia (Cardiac disorders) | 12 (15)
Exacerbation of heart failure (Cardiac disorders) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Inappropriate High Voltage therapy (Injury, poisoning and procedural complications) | 7 (7)
Inappropriate low voltage therapy (Injury, poisoning and procedural complications) | 4 (4)
Lead dislodgement or migration (Injury, poisoning and procedural complications) | 3 (3)
Other cardiovascular (Cardiac disorders) | 11 (13)
Other non cardiovascular (General disorders) | 14 (15)
device oversensing (Injury, poisoning and procedural complications) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Device threshold elevation (Injury, poisoning and procedural complications) | 2 (2)
Vein thrombosis (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Additional investigation into ST segment changes in advance of VT/VF, including their association to confirmed ischemic events, is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less